CLINICAL TRIAL: NCT05557201
Title: Cohort of Patients Presenting Unexplained Recurrent Miscarriages and Identification of Early Miscarriage Recidivism Factors
Acronym: FALCO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220747; IDRCB 2022-A00273-40 (Other: ANSM)
Record Dates: First submitted 2022-09-08; First posted 2022-09-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Miscarriage; Early Pregnancy Loss
Keywords: Miscarriage; Prognostic factors; Biological collection; recurrent early pregnancy losses; repeated implantation failure
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Miscarriage: Patients with recurrent early pregnancy losses (at least 3 fetal losses before 14 weeks of amenorrhea) and/or recurrent implantation failures (at least 3 failures).

SUMMARY:
About 1 to 3% of women of childbearing age suffer repeated early spontaneous miscarriages (RCF) defined by at least 3 fetal losses before 14 weeks of gestation. RCFs may be linked to parental chromosomal abnormalities, congenital or acquired uterine abnormalities, hormonal causes (e.g. type 1 and 2 diabetes, ovarian failure), infectious etiology, constitutional or acquired thrombophilia or sickle cell disease.

The presence of antiphospholipid antibodies, antithyroid and anti-transglutaminase antibodies in approximately 10% of cases suggests an autoimmune origin for these fetal losses. The role of other antibodies, in particular non-conventional antiphospholipid antibodies, remains to be established. Indeed half of RCF cases are thought to be due to an immunological dysregulation of the mother leading to a decrease in tolerance to the fetus. Several studies have shown immune abnormalities, such as an imbalance of pro and anti-inflammatory cytokines, an increase in cytotoxic cells and a defect in regulatory cells in the blood of patients. The assessment of these immune abnormalities is not currently performed routinely in France in women presenting with recurrent early miscarriages. When one of these known causes is excluded, it is unexplained RCF which represents 50% of RCF. Over half of these women with RCF may be linked to aneuploidies and primary spontaneous recurrent abortions. Assessing the degree of aneuploidy and the genetic origin of foetal losses remains difficult to date, as examination of the miscarriage product is rarely available, due to the spontaneous nature of the loss.

An implantation failure (IF) is defined as the absence of pregnancy following the transfer of a good-quality embryo into the uterine cavity. These implantation failures can be due to embryonic factors, maternal factors, or caused by inappropriate stimulation and/or difficult transfers. In the literature, recurrent implantation failure (RIF) is defined as the absence of pregnancy after 3 attempts of transferring good-quality embryos, taking maternal age into account Setting up a prospective cohort of patients with RFC is an essential step in exploring the aetiological factors of RCF and in order to enable better treatment.

DETAILED DESCRIPTION:
The study population will be followed as part of routine care, in the same way as all patients presenting with RPL, in internal medicine or obstetrics-gynecology.

On the day of inclusion, the patient's medical history will be reviewed (demographic data, lifestyle factors, medical and obstetric-gynecologic history, biological tests performed).

Data for each of the patient's pregnancies will also be collected (date of pregnancy onset, type of pregnancy, pregnancy outcome, treatments taken during pregnancy, maternal/fetal complications during pregnancy).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years
* Patients who have had 3 (or more) early pregnancy losses occurring before 14 weeks of amenorrhea and/or at least 3 implantation failures.
* Patients who have been informed and have not objected to participating in the study.
* Patients covered by a social security system.

Exclusion Criteria:

* patients who do not agree the use of their data
* Patients on AME
* Patients under legal protection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with recurrent early pregnancy losses (at least 3 fetal losses before 14 weeks of amenorrhea) and/or recurrent implantation failures (at least 3 failures).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
To build a cohort of patients in order to describe clinical characteristics, tests carried out and medical care of patients presenting spontaneous recurrent miscarriages | through study completion, an average of 5 years
  Description of the clinical and biological characteristics of patients with recurrent early pregnancy losses and/or recurrent implantation failures

SECONDARY OUTCOMES:
To describe the recurrence rate of repeated early pregnancy loss | Through study completion, an average of 5 years
  Proportion of recurrence of early pregnancy loss (EPL) over the entire duration of the study: according to the number of previous early pregnancy losses; according to abnormalities found in the etiological work-up; according to age at onset, associated infertility, type of pregnancy loss with or without live children, and according to the different treatments used
To describe the recurrence rate of repeated implantation failure | Through study completion, an average of 5 years
  Proportion of recurrence of RIF over the entire duration of the study: according to the number of previous implantation failures, according to abnormalities found in the etiological work-up, according to age at onset, associated infertility, and according to the different treatments used
To compare the efficacy of immunomodulatory drugs (corticosteroids, hydroxycholoroquin, Intravenous Immunoglobulin Therapy, intralipids, biotherapies) | through study completion, an average of 5 years
  Description of the efficacy of the various drugs : number of full term pregnancies
To evaluate the psychological state of patients and the impact on pregnancy | through study completion, an average of 5 years
  Evaluation of the patients' lifestyle using the Baecke questionnaire and medical interrogation.
to evaluate patients' lifestyle and the impact on pregnancy | evaluation of the patients' lifestyle using the Baecke questionnaire and medical interrogation.
  through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Arsene MEKINIAN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Internal medicine department, hospital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dernoncourt A, Hedhli K, Abisror N, Cheloufi M, Cohen J, Kolanska K, McAvoy C, Selleret L, Ballot E, Mathieu d'Argent E, Chabbert Buffet N, Fain O, Kayem G, Mekinian A. Hydroxychloroquine in recurrent pregnancy loss: data from a French prospective multicenter registry. Hum Reprod. 2024 Sep 1;39(9):1934-1941. doi: 10.1093/humrep/deae146. PMID 38942601